CLINICAL TRIAL: NCT02885896
Title: Cluster-randomized Controlled Study Evaluating the Impact of a Call Center Providing Standardized Pediatric Advices Based on the Number of Unscheduled and Medically Unjustified Consultations
Brief Title: Assessing the Impact of a Call Center Providing Standardized Pediatric Advice (PLATEL-EVAL)
Acronym: PLATEL-EVAL
Status: Withdrawn | Type: Observational
Why Stopped: Principal investigator left the Hospices Civils de Lyon and has not been replaced
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D50849
Record Dates: First submitted 2016-08-23; First posted 2016-09-01 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Emergency Pediatric Care
Keywords: Call center; nurses; pediatrics; standardized messages; family counseling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental period (active platform): During the experimental period, the eligible calls will be transferred to the platform by SAMU regulator doctors, and callers will be subject to health advice by specially trained nurses. The nurse conduct the call by holding the conversation guide, giving advice for a home care, answering questions from the circle (caller, family,..) and ensuring the proper understanding of these tips. An information leaflet for the theme of the call will be sent in the days following the call to the caller of the experimental group having given their consent.
- Control period (inactive platform): During the control periods, the call center will not be active, eligible calls can not receive advice from nurses, but will be subject to the usual care: the regulator doctor will treat the call as its current practice.

SUMMARY:
In order to show that tailored pediatric counselling by telephone can reduce the number of unscheduled and medically unjustified physicians visits in emergency structures, a randomized controlled study is conducted. It compares the proportion of cases which used the emergency services or unscheduled consultation according to whether they received (or not) nurses' telephone advices from the platform. Indeed, our hypothesis is that the presence of nurses responding at the Reception and Control Calls Center inside the Emergency Medical Services (in french : Service d'Aide Médicale d'Urgence SAMU) - whose role is to deliver appropriate advice to people calling for benign pathologies they see as urgent and to answer questions following specific recommendations - will reduce the number of unplanned and medically unjustified consultations in medical emergency structures.

This platform was set-up in order to show it may be a solution in response to the growing demand for pediatric care from the population, helping to reduce overcrowding in emergency care facilities. Indeed, promoting home care or only if necessary scheduled consultation reinforces the conduct to have when facing a pathology from their child. It will also help by reducing unjustified use of emergency structures, improving not only the users' reception conditions who actually require support in these structures with less waiting time, but also the working conditions for employees who perform there.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are different depending on the subject concerned, for reasons related to risk factors of pediatric diseases. They are audited by the regulator doctor (who has a fact sheet) and are controlled by the nurse of the platform.
* For fever theme, a call is eligible if the child is older than 3 months and under 6 years old, and has had a fever for less than 48 hours.
* For the theme diarrhea, a call is eligible if the child in question is aged from 12 months to 3 years, and has had diarrhea. Fever and vomiting are not exclusion criteria.
* For the theme breathing difficulty, a call is eligible if the child in question is aged from 3 months to 3 years, has experienced discomfort breathing and has shown no fever. Stuffy nose, runny nose and cough are not exclusion criteria.
* For the theme fall with head shock, a call is eligible if the child concerned is a toddler and until the age of 12.
* For the theme crying infant, a call is eligible if the child in question is aged 0-4 months and has been crying. Fever is an exclusion criterion.

Exclusion Criteria:

* Refusal of participation or refusal to be reminded to 7 days,
* Children with impaired general condition and / or behavior change during the call,
* Situation requiring medical attention without delay,
* Lack of understanding of the caller

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children whom parents call the center 15 for pediatric advice
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Number of unscheduled consultations | up to 7 days after inclusion
  The main objective of the study is to compare the number of unscheduled consultations within 7 days following inclusion, i.e. the call at Centre15 (reception and regulation calls center) between the sample with access to telephone advice and the one who received the usual care (control group) . Our assumption is that the number of appeals for emergency medical services will be lower in the group that received advice from the platform than in the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Hcl-Ghe-Epicime, Bron, France